CLINICAL TRIAL: NCT06763341
Title: A Phase 1 Study of AOH1996 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24727; NCI-2024-10209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24727 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Specimen Handling; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort I (AOH1996) (Experimental): Patients receive AOH1996 PO BID on days 1 - 28 of each cycle. Cycles repeat every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients that attain a CR/CRh/CRi with transfusion independence (TI) by the end of cycle 2 continue cycles every 28 days for up to 12 total cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow aspiration and blood sample collection throughout the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: PCNA Inhibitor AOH1996; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: PCNA Inhibitor AOH1996 — Given PO
  Other Names: AOH1996; Proliferating Cell Nuclear Antigen Inhibitor AOH1996; AOH
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase 1 trial tests safety, side effects, and best dose of AOH1996 for the treatment of patients with acute myeloid leukemia (AML) that has come back after a period of improvement (relapsed) or AML that has not responded to previous treatment (refractory). AOH1996 is in a class of medications called PCNA inhibitors. It inhibits cancer growth and induces deoxyribonucleic acid (DNA) damage. This may help keep cancer cells from growing and damage cancer cell DNA. Giving AOH1996 may be safe, tolerable and/or effective in treating patients with AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of AOH1996 in patients with relapsed/refractory (R/R) acute myeloid leukemia (AML).

II. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of AOH1996.

SECONDARY OBJECTIVES:

I. Evaluate the anti-leukemic activity, as assessed by complete remission (CR) rate at the end of cycles 1 and 2.

II. Evaluate the anti-leukemic activity, as assessed by overall response rate ([ORR]: CR+CR with incomplete hematologic recovery rate [CRi]+CR with partial hematologic recovery [CRh]+morphologic leukemia-free state [MLFS] + partial remission [PR]) at the end of cycles 1 and 2.

III. Evaluate the anti-leukemic activity, as assessed by complete remission (CR), overall response (ORR: CR+CRi+CRh+PR) and minimal residual disease (MRD)- rate and duration over the study period.

IV. Evaluate transfusion independence (TI). V. Estimate overall survival (OS) rate, progression-free survival (PFS) and duration of response (DOR) rate at 6 months and 1 year.

VI. Describe the plasma pharmacokinetics (PK) of AOH1996 alone.

EXPLORATORY OBJECTIVES:

I. Determine biomarkers that may be predictive of AOH1996 activity. II. Study the impact of AOH1996 on altered mitochondrial metabolism and dynamics.

III. Determine pharmacodynamics (PD) parameters (alteration of OPA1) of AOH1996.

IV. Estimate leukemia stem cell burden in bone marrow pre-, post-therapy. OUTLINE: This is a dose-escalation study of AOH1996.

COHORT I: Patients receive AOH1996 orally (PO) twice daily (BID) on days 1 - 28 of each cycle. Cycles repeat every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients that attain a CR/CRh/CRi with transfusion independence (TI) by the end of cycle 2 continue cycles every 28 days for up to 12 total cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow aspiration and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 30 days and up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy > 3 months
* Patients with histologically confirmed AML, according to International Consensus Classification (ICC) or World Health Organization (WHO) criteria, with refractory/relapsed (R/R) disease who have failed treatment with, or are ineligible for, available therapies known to be effective for treatment of their AML

  * Patients with extramedullary disease may be included if they also have marrow involvement
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Ability to swallow pills
* White blood cell (WBC) ≤ 25 x 10^9/L prior to initiation of study therapy. Cytoreduction with hydroxyurea prior to treatment and/or during cycle 1 may be required (within 14 days prior to day 1 of protocol therapy)
* Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 3.0 x ULN (within 14 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 3.0 x ULN (within 14 days prior to day 1 of protocol therapy)
* Creatinine clearance of ≥ 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 14 days prior to day 1 of protocol therapy)
* International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN (within 14 days prior to day 1 of protocol therapy)
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (within 14 days prior to day 1 of protocol therapy)
* Corrected QT interval (QTc)F ≤ 480 ms based on Fridericia's formula

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 14 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control (nonhormonal) or abstain from heterosexual activity for the course of the study through at least 2 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Hematopoietic stem cell transplant within 100 days prior to day 1 of protocol therapy. Patients who have stopped calcineurin inhibitors (CNI) must be off CNIs for at least 2 weeks prior to day 1 of protocol therapy
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 14 days prior to day 1 of protocol therapy with the following exception of hydroxyurea which is allowed prior to treatment and through cycle 1 for control of rapidly progressing leukemia
* Strong inducers or strong inhibitors of CYP enzymes (e.g., 1A2, 2B6, 2C8, 2C9, 2C19, and 3A4), other than azole antifungals with CYP3A4 inhibition potential, or drug transporters (e.g., organic anions [OATP1B1/1B3], BCRP, P-gp, organic cations [OCT1, OCT2, OCT3], MATE1 or MATE2K), or sensitive substrates of these CYPs or drug transporters, within 4-5 half-lives or 14 days prior to the first dose of study drug, whichever is longer.
* Foods/supplements that are strong inhibitors or strong or moderate inducers of CYP3A (such as St. John's wort) within 3 days prior to initiation of and during study treatment
* Systemic steroid therapy > 10 mg/day (≤ 10mg/day prednisone equivalent ok) or any other form of immunosuppressive medication within 14 days. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted
* Must not have received or planning to receive live vaccine while being on study or 4 weeks before and after completion of treatment
* Patients with blast phase chronic myeloid leukemia (CML)
* Patients with translocation (t)(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Active central nervous system (CNS) disease
* Active graft versus (vs) host disease (GVHD)
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * Uncontrolled atrial fibrillation or hypertension
* No measurable disease in the bone marrow
* Gastrointestinal disorder that interferes with oral drug absorption such as malabsorption syndrome
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Uncontrolled active infection
* Clinically significant uncontrolled illness
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2027-01-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | During cycle 1 (Cycle length = 28 days)
  Will evaluate for DLTs in patients that receive at least 75% of the planned dose(s) of AOH1996 per dose level assignment. In-evaluable subjects will be replaced. Will grade toxicity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Incidence of adverse events | Up to 2 years
  Will evaluate toxicity in patients that receive any AOH1996. Will grade toxicity according to the NCI CTCAE v5.0. Will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Response | Up to 1 year
  Will evaluate in all eligible patients with a baseline assessment who start therapy (i.e., receiving at least one dose of a AOH1996). These patients will be considered in the primary analysis of response rate as the denominator, with number of responders in the numerator. Patients will have their response classified according European LeukemiaNet criteria of Dohner and others (2022). Response rates will also be explored based on number/type of prior therapy(ies).
Minimal residual disease (MRD) status | Up to 1 year
  Will be determined by conventional care flow cytometry assay performed locally using a 0.01% blast threshold for positivity. Will report MRD over the study period using both descriptive statistics and graphical methods.
Complete remission (CR) | From start of treatment to attainment of CR/CR with incomplete hematologic recovery rate (CRi)/CR with partial hematologic recovery (CRh), assessed up to 1 year
  Will evaluate time to CR. Rates and 95% Clopper-Pearson binomial confidence interval will be calculated for the complete remission rate (CR/CRi/CRh). Response rates will also be explored based on number/type of prior therapy(ies).
First response | From start of treatment to attainment of first documented CR/CRi/CRh/morphologic leukemia-free state/partial response, assessed up to 1 year
  Will evaluate time to first response.
Duration of response (DOR) | Time interval from the date of first documented response (CR+CRi+CRh) to the date of documented disease relapse or death whichever occurs first, assessed up to 2 years
  Will evaluate DOR. Will be estimated using the product-limit method of Kaplan and Meier.
Overall survival (OS) | Time interval from start of study treatment to the date of death from any cause, assessed up to 2 years
  Will evaluate OS. OS will be censored at last follow-up if patients are known to be alive. Will be estimated using the product-limit method of Kaplan and Meier.
Progression-free survival (PFS) | Time interval from start of study treatment to the date of first documented disease relapse/progression or death from any cause, whichever occurs first, assessed up to 2 years
  Will evaluate PFS. PFS will be censored at last follow-up if patients are alive and relapse/progression-free. Will be estimated using the product-limit method of Kaplan and Meier.
AOH1996 in plasma | 0-2 hours pre-dose and 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, and 24 hours post-dose on days 1 and 8 of cycle 1 (Cycle length= 28 days) and pre-dose and 1-3 h post-dose of the morning doses on day 1 of cycles 2-12
  Will evaluate levels of AOH1996 in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Blackmon, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States